CLINICAL TRIAL: NCT03823677
Title: Analysis of Protein and Emotional Alterations During and After Hypobaric Hypoxia
Acronym: DRU-EMO-K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Principal Investigator, Jochen Hinkelbein, Clinical Professor, Universitätsklinikum Köln
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DRU-EMO-KOELN
Record Dates: First submitted 2019-01-07; First posted 2019-01-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Hypoxia, Altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Intervention Model Description: 15 different Groups are analysed: control Group, 5000ft Group, 8000 ft Group, 10000ft Group and 15000ft Group - all for 15, 30, and 60 minutes.
Who Masked: Participant
Masking Description: volunteers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- control group 15 (No Intervention): Protein expression and emotional test
  15 minutes normoxia
  Interventions:
  Blood drawing 1 Minute before and 1 Minute after the pressure chamber Phase for Proteomic profiling with 2D-gels
  Emotional tests (tears, stroop, mood) during the pressure chamber phase
- control group 30 (No Intervention): 30 minutes normoxia
  Interventions:
  Blood drawing 1 Minute before and 1 Minute after the pressure chamber Phase for Proteomic profiling with 2D-gels
  Emotional tests (tears, stroop, mood) during the pressure chamber phase
- control group 60 (No Intervention): 60 minutes normoxia
  Interventions:
  Blood drawing 1 Minute before and 1 Minute after the pressure chamber Phase for Proteomic profiling with 2D-gels
  Emotional tests (tears, stroop, mood) during the pressure chamber phase
- hypoxia 5000ft group 15 (Experimental): Intervention: 15 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 5000ft group 30 (Experimental): Intervention: 30 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 5000ft group 60 (Experimental): Intervention: 60 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 8000ft group 15 (Experimental): Intervention: 15 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 8000ft group 30 (Experimental): Intervention: 30 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 8000ft group 60 (Experimental): Intervention: 60 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 10000ft group 15 (Experimental): Intervention: 15 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 10000ft group 30 (Experimental): Intervention: 30 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 10000ft group 60 (Experimental): Intervention: 60 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 15000ft group 15 (Experimental): Intervention: 15 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 15000ft group 30 (Experimental): Intervention: 30 minutes hypoxia
  Interventions: Procedure: Hypoxia
- hypoxia 15000ft group 60 (Experimental): Intervention: 60 minutes hypoxia
  Interventions: Procedure: Hypoxia

INTERVENTIONS:
Procedure: Hypoxia — hypoxia
  Arms: hypoxia 10000ft group 15; hypoxia 10000ft group 30; hypoxia 10000ft group 60; hypoxia 15000ft group 15; hypoxia 15000ft group 30; hypoxia 15000ft group 60; hypoxia 5000ft group 15; hypoxia 5000ft group 30; hypoxia 5000ft group 60; hypoxia 8000ft group 15; hypoxia 8000ft group 30; hypoxia 8000ft group 60

SUMMARY:
This study analyses both Protein Expression and emotional alterations during hypobaric hypoxia in volunteers of different groups.

DETAILED DESCRIPTION:
This study analyses both Protein Expression and emotional alterations during hypobaric hypoxia in volunteers of different groups.

15 different Groups are analysed: control Group, 5000ft Group, 8000 ft Group, 10000ft Group and 15000ft Group - all for 15, 30, and 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Helathy

Exclusion Criteria:

* Ear problems

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Protein Expression before hypoxia | Measurement immediately 1 minute before of hypoxia/experiment
  proteomic profiling of Serum by 2D-gels. All Proteins present in the sample will be identified by proteomics
Protein Expression after hypoxia | Measurement immediately and at termination (i.e., 1 minute after) of hypoxia/experiment
  proteomic profiling of Serum by 2D-gels. All Proteins present in the sample will be identified by proteomics
Emotional assessment tears | Measurement starts immediately with hypoxia in the pressure chamber. duration 10 minutes
  Emotional tears test
Emotional assessment | Measurement in the pressure chamber after tears test (i.e. 10 minutes after start). duration 10 minutes
  Emotional stroop test; Williams, J. M. G., Mathews, A., & MacLeod, C. (1996). The emotional Stroop task and psychopathology. Psychological Bulletin, 120, 3-24.
Emotional assessment mood | Measurement in the pressure chamber after stroop test (i.e. 20 minutes after start). duration 10 minutes
  Emotional mood test, POMS mood score. Shukitt-Hale, B., Banderet, L.E., & Lieberman, H.R. (1998). Elevation-dependent symptom, mood, and performance changes produced by exposure to hypobaric hypoxia, The International Journal of Aviation Psychology, 8, 319-334,

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Hinkelbein, Study Chair — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No